CLINICAL TRIAL: NCT01166750
Title: Jointstrong Intervention for Juvenile Arthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Rapoff, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Michael Rapoff, Ph.D., Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11154
Record Dates: First submitted 2010-07-19; First posted 2010-07-21 (Estimated); Results first posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Juvenile Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — CD-ROM

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CD-ROM-treatment (Experimental)
  Interventions: Behavioral: CD-ROM
- Wait-list Control Group (Active Comparator)
  Interventions: Behavioral: Wait-list Control Group

INTERVENTIONS:
Behavioral: CD-ROM — Treatment Group will continue to follow their treating rheumatologist's recommendations and prescriptions. The program will contain information on the multiple components of pain (the "pain puzzle") as a treatment rationale and will then teach children to use cognitive-behavioral techniques for pain management. The information will be presented via visual displays, narration, and interactive menus. Children will be able to navigate through the different lessons at their own pace and will be required to take simple quizzes to assess their learning. Various passwords and homework assignments are embedded within the program to ensure that children are going through the material.
  Arms: CD-ROM-treatment
Behavioral: Wait-list Control Group — Children in the control group will continue to follow recommendations and prescriptions by their treating rheumatologist. After an 8-week wait-list control condition that involves measurement phases identical to those of the Jointstrong Treatment Group but no Jointstrong treatment, the children in the control group will enter the Jointstrong program and will then have the same immediate post-treatment measures that the Treatment Group received. The Control Group will not, however, have the Treatment Group's 12-week follow-up phase.
  Arms: Wait-list Control Group

SUMMARY:
This study is a randomized wait-list controlled trial with repeated measures. There will be two groups: (1) standard medical care (wait-list control), and (2) standard medical care plus the adjunctive Jointstrong pain coping skills CD-ROM program (treatment). The study will have four phases: Pre-intervention Baseline (2 weeks); Intervention (4 weeks); immediate post-intervention follow up (2 weeks); and 12-week post-intervention follow up (2 weeks). The purpose of this study is to determine if using a CD-ROM program for juvenile arthritis can help children learn how to improve their symptoms on their own and reduce the frequency of symptoms.

DETAILED DESCRIPTION:
If your child is eligible and decides to participate in this study, this participation will last approximately eight weeks. Please refer to the table at the end of this consent form.

Your child's participation in this study will involve the completion of daily questionnaires during a one-week baseline period and a one-week follow-up period. These questionnaires will contain various questions about your child's arthritis and his/her ability to do various activities. The questionnaires will take approximately 15-30 minutes each week to complete.

Your child will be randomly assigned to complete one of two CD-ROM programs. One of the CD-ROM programs is a "control" program that contains educational information about arthritis and medical treatments and the other is the "treatment" program and contains the same educational information as the control program plus information on behavioral strategies for controlling symptoms of arthritis. Your child's participation in this study will involve working through one of these CD-ROM programs over a one-month period. Your child will also continue to receive medical treatment from the rheumatologist treating your child for arthritis. The CD-ROM programs involve working through developmentally appropriate lessons on the nature of arthritis and how to treat it. The CD-ROM programs are divided into weekly "modules" and are designed to be completed within four weeks. Lessons take an average of 15 minutes to complete (plus "homework"), and there is an average of 4 lessons to complete each week.

Your participation in this study will involve the completion of questionnaires and helping your child understand any parts of the study that he or she does not understand.

ELIGIBILITY:
Inclusion Criteria. Patients recruited for this study will meet the following inclusion criteria: (a) are 8-12 years of age; (b) have a diagnosis of JA by a pediatric rheumatologist using established criteria, and (c) have JA-related (joint) pain occurring on an average of at least once per week by patient report [9]. Participants in the age range 8-12 years will be recruited because the intervention will be tailored to children (future studies will involve creating and testing a version of Jointstrong for adolescents). Although access to a home computer with a CD-ROM drive is required for the study, this will not be an inclusion criterion, and we expect the lack of access will be rare, as our pilot data on 37 children with headaches found that only 2% (1 child) did not have adequate home computer access [15]. So as not to exclude the few children without access who otherwise qualify for the study, we will lend laptop computers to these children. All children meeting symptom inclusion criteria will therefore be able to use the adjunctive CD-ROM programs in a home setting.

Exclusion Criteria. Patients will be excluded from the study if (a) their parents or rheumatologist report they have been diagnosed with a mental health condition or they are receiving concurrent psychotherapy; or (b) their 14-day baseline pain diaries indicate they have pain, on average, less than one day per week; or (c) they do not speak English.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2009-04; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rapoff, Ph D, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University Of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment were from April 2009 to May 2011.
Pre-assignment Details: Twelve subjects were not randomized to groups, 2 due to infrequent pain, 2 moved or phone was disconnected, 6 would not return phone calls, and 2 dropped out as they were too busy.
Groups:
- CD-ROM-treatment: CD-ROM : Treatment Group will continue to follow their treating rheumatologist's recommendations and prescriptions. The program will contain information on the multiple components of pain (the "pain puzzle") as a treatment rationale and will then teach children to use cognitive-behavioral techniques for pain management. The information will be presented via visual displays, narration, and interactive menus. Children will be able to navigate through the different lessons at their own pace and will be required to take simple quizzes to assess their learning. Various passwords and homework assignments are embedded within the program to ensure that children are going through the material.
- Wait-list Control Group: Wait-list Control Group : Children in the control group will continue to follow recommendations and prescriptions by their treating rheumatologist. After an 8-week wait-list control condition that involves measurement phases identical to those of the Jointstrong Treatment Group but no Jointstrong treatment, the children in the control group will enter the Jointstrong program and will then have the same immediate post-treatment measures that the Treatment Group received. The Control Group will not, however, have the Treatment Group's 12-week follow-up phase.
Period: Overall Study
Arm/Group | CD-ROM-treatment | Wait-list Control Group
Started | 10 | 13
Completed | 9 | 13
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD-ROM-treatment | Wait-list Control Group | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10 | 13 | 23
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 10.3 (1.2) | 10.6 (1.6) | 10.5 (1.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 9 | 18
  Male | 1 | 4 | 5
Region of Enrollment [Number; unit: participants]
  United States | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: Pain
Description: Pain intensity on a 0 to 10 visual analog scale with 0 being no pain and 10 being worst possible pain.
Time Frame: weekly for 12 weeks
Population: They were the ones still remaining at the end of the study.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- CD-ROM Treatment: Jointstrong
Arm/Group | CD-ROM Treatment | Wait-List Control Group
Number analyzed (Participants) | 9 | 13
units on a scale | 4.3 (1.8) | 5.7 (3.3)

2. Secondary Outcome: Mood and Stress
Time Frame: weekly for 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Quality of Life
Time Frame: weekly for 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | CD-ROM-treatment | Wait-list Control Group
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/13
Other Adverse Events (participants affected / at risk) | 0/9 | 0/13

LIMITATIONS AND CAVEATS:
It was difficult to find subjects with pain resulting in significantly fewer subjects entered in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes